CLINICAL TRIAL: NCT05805618
Title: A Single-center, Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Safety and Immunogenicity of Recombinant Norovirus Hexavalent Vaccine in Healthy Subjects Aged 18-59 Years
Brief Title: Evaluation of Recombinant Norovirus Hexavalent Vaccine in Healthy Subjects
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Syneos Health (Other)
Collaborators: Chengdu Kanghua Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: KH-CT-002-01
Record Dates: First submitted 2023-02-23; First posted 2023-04-10 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KH002 (Experimental): at low dose,150 mg(Cohort 1 ), 20 subjects are dosed Vaccine as experimental at high dose,300mg (Cohort 2), 20 subjects are dosed Vaccine as experimental
  Interventions: Biological: Recombinant Norovirus Hexavalent Vaccine
- matching placebo (Placebo Comparator): at low dose,150 mg(Cohort 1 ), 10 subjects are dosed placebo at high dose, 300mg(Cohort 2),10 subjects are dosed placebo
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Biological: Recombinant Norovirus Hexavalent Vaccine — To prevent acute gastroenteritis caused by norovirus of genotypes GI.1, GII.2, GII.3, GII.4, GII.6, and GII.17
  Other Names: KH002
  Arms: KH002
Other: Matching Placebo — matching placebo for Recombinant Norovirus Hexavalent Vaccine / KH002
  Arms: matching placebo

SUMMARY:
To evaluate the safety and immunogenicity of different dose levels of the Recombinant Norovirus Hexavalent Vaccine in healthy subjects aged 18-59 years given three doses of the vaccine at 28-day intervals.

DETAILED DESCRIPTION:
It is planned to enroll healthy subjects and adopt a 3-dose vaccination schedule (day 0 to day 56) of intramuscular injections of study vaccines in the deltoid muscle of the upper arm of subjects on day 0, day 28 and day 56, respectively. The subjects will sequentially enter into the low and high dose groups by stages, with approximately 30 subjects in each group (test group:control group = 2:1) and approximately up to 60 subjects in total. At least half of the subjects are Chinese in the two cohorts respectively

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-59 years (inclusive);
2. Subjects with a body mass index ( 18 kg/m2 and 35 kg/m2;
3. Capable and willing to give informed consent prior to any study-specific activities/procedures;
4. Subjects who are able to comply with the requirements of the clinical study protocol to complete the study;
5. Subjects who haven't been vaccinated or haven't plan to be vaccinated with other vaccines (including live attenuated vaccines, non-live vaccines, and novel coronavirus vaccines) within 14 days before the first dose of study vaccines;
6. Subjects who are clinically determined to be healthy by the investigator after being inquired about their medical history and relevant physical examinations;
7. Female subjects who are not breastfeeding; all subjects who have no childbearing plan or sperm/egg donation plan from ICF signing to 6 months after the completion of the vaccination series and agree to take effective contraceptive measures (See the appendix 3) from 4 weeks prior to the first dose to 6 months after the completion of the vaccination series.

Exclusion criteria for the first vaccination dose

1. Subjects with positive COVID-19 test by PCR for nasopharyngeal or oropharyngeal swabs (nasopharyngeal swabs are preferred) on the day of the first dose vaccination;
2. Subjects who have previously participated in a clinical study of any type of norovirus vaccines within the past year before enrollment in this study;
3. Subjects with a history of chronic gastrointestinal disorder or having gastroenteritis that required treatment (for example, seek medical advice, etc.) within the past year before screening; or subjects have diarrhea, vomiting, or other digestive system conditions before 2 weeks of the first dose vaccination;
4. Subjects have cancer or have a history of cancer within 5 years before screening;
5. Subjects with the following conditions: (1) serious congenital malformations, serious developmental disorders, serious genetic defects, serious malnutritions, etc.; (2) thrombocytopenia, coagulation disorder or receipt of anticoagulant therapy, and other contraindications to intramuscular injections; (3) congenital or acquired immunodeficiency or receipt of immunosuppressant therapy (excluding topical treatment, surface treatment for acute non-complicated dermatitis, spray treatment for allergic rhinitis, ICS use for asthma treatmen, etc.) within 6 months; (4) history of infectious diseases, such as tuberculosis; (5) history or family history of convulsions, epilepsy, encephalopathy; (6) asplenia, functional asplenia, and asplenia or splenectomy due to any cause; (7) serious cardiovascular diseases (pulmonary heart disease and pulmonary edema), serious liver and kidney diseases, type I diabetes, celiac disease, autoimmune diseases, etc.; (8) use of medications within the timeframes specified in Section 6.5.2 ;
6. Subjects with a clinicallly significant history of serious hypersensitivity to any component of study vaccines, including adjuvant components and yeast, such as allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, and local allergic necrotic reaction (Arthus reaction); a history of serious adverse vaccine or drug reactions, such as allergy, urticaria, skin eczema(small, local rashes on a single body part are permitted), dyspnea, and angioedema;
7. Subjects with abnormal and clinically significant results of laboratory tests at the discretion of Investigator, such as hematology, serum chemistry, and urinalysis;
8. Subjects with abnormal and clinically significant ECG results up to the Investigator's discretion at screening;
9. Females of childbearing potential with positive serum pregnancy test results;
10. Subjects who are positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) antibody, or anti-treponema pallidum (anti-TP) antibody at screening;
11. Subjects with hypertension (systolic blood pressure 140 mmHg and/or diastolic blood pressure 90 mmHg) or hypotension (systolic blood pressure < 90 mmHg and/or diastolic blood pressure 40 mmHg) (regardless of medication use) in the physical examination before enrollment;
12. Subjects with fever (oral temperature ≥ 37.5 °C) on the day of vaccination with study vaccines or within 72 h before vaccination;
13. Subjects who have donated blood or lost blood (≥ 400 mL) or received blood transfusion or used blood products within 30 days before signing the ICF or plan to donate blood during the study(from the first vaccination dose to 3 months after the completion of the vaccination series);
14. Subjects who have undergone surgery within 3 months before signing the ICF or plan to undergo surgery (including cosmetic surgery, dental surgery, and oral surgery(excluding tooth filling, protaper and tooth extraction)) during the study (from the first vaccination dose to 3 months after the completion of the vaccination series);
15. Smoking more than 10 cigarettes per week within 3 months prior to screening;
16. History of alcohol abuse within 1 year prior to screening, or regular use of alcohol within 6 months prior to screening that exceeds 14 units of alcohol per week (1 unit = 375 mL of beer 3.5%, 100 mL of wine 13.5%, or 30 mL of spirit 40%);
17. History of drug abuse within 1 year prior to screening, or recreational use of soft drugs (such as marijuana) or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, codeine and amphetamine derivatives) within 1 month prior to screening;
18. Subjects with positive tests for drugs of abuse (including Amphetamines (AMP), Methamphetamines (MET), Methadone (MTD), Barbiturates (BAR), Benzodiazepines (BZO), Cocaine (COC), Opiates (OPI), Methyl enedioxy methamphetamine (MDMA) , Phencyclidine (PCP), Tetrahydrocannabinol (THC)) and alcohol breath test;
19. Subjects with tattoos, scars or skin defects covering the deltoid muscle who are not suitable to participate in the study up to the investigator's discretion;
20. Subjects who cannot tolerate venipuncture or have a history of fear of needles or hemophobia;
21. Subjects who are not suitable to participate in the study as determined by the investigator .

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of solicited AEs within 7 days after each vaccination dose. | 7 Days
  Safety will be assessed through 7 days after vaccination (including the day of vaccination) via collection of solicited AEs. The solicited AEs include local AEs (injection site: pain,tenderness， induration,swelling,erythema,pruritus)and systemic AEs (Headache, Fatigue,Myalgia,Arthralgia,Vomiting, Diarrhea, Fever).
Incidence of unsolicited AEs within 28 days after each vaccination dose | 28 Days
  Unsolicited AEs are AEs other than those designated as solicited AEs, and also include eponymous solicited AEs that occur after the solicitation period. Unsolicited AEs mainly include any AEs that have been reported by the subjects, learned from interrogation or observed by the investigator during the study visits, or discovered during review of medical records or original files. the incidence of unsolicited AEs within 28 days after each dose of the study vaccine will be calculated.
Incidence of AEs related to serum chemistry, hematology, and urinalysis parameters in all subjects on day 4 after each vaccination dose and on day 14, day 42 after the first dose | 42 days
  The number of participants with any markedly abnormal standard safety laboratory values (serum chemistry,hematology or urinalysis) collected.
SAE, MAAE in all subjects within 12 months after the completion of the vaccination series. | 12 Months
  The subjects will also be monitored for SAEs, MAAEs from the first dose to 12 months after the completion of the vaccination series.

SECONDARY OUTCOMES:
GMT of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP HBGA (BT50) | 12 Months
  GMT is geometric mean titer. HBGA is Histo-blood group antigen. Predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination (up to Day 421)
GMFR of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP HBGA | 12 Months
  GMFR is geometric mean fold rise. Predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination (up to Day 421)
SCR of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP HBGA | 12 Months
  SCR is Seroconversion rate. Seroconversion is defined as: For the subject whose antibody titer is below the lower limit of quantification before vaccination, the antibody titer is increased to the lower limit of quantification or above after vaccination; for the subject whose antibody titer is at the lower limit of quantification or above before vaccination, the antibody titer is increased at least 4-fold after vaccination. Predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination
GMT of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP Pan-Ig | 12 Months
  predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination
GMFR of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP Pan-Ig | 12 Months
  Predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination
SCR of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP Pan-Ig | 12 Months
  Predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination
GMT of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP IgA | 12 Months
  Predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination
GMFR of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP IgA | 12 Months
  Predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination
SCR of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP IgA | 12 Months
  Predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination
GMT of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP IgG | 12 Months
  Predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination
GMFR of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP IgG | 12 Months
  predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination
SCR of Serum Anti-norovirus GI.1 and GII.2, GII.3, GII.4, GII.6, GII.17 VLP IgG | 12 Months
  Predose 0 and 7, 14, 28 days after the first and second dose, and 7, 14, 28 days, 3, 6, 12 months after completion of full vaccination
Norovirus-specific T-cell IFN-γ,IL-2, IL-4 and IL-10 levels In the high dose group. | 28 Days
  Predose 0 and 7, 28 days after completion of full vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Kristi McLendon, Dr, Principal Investigator — Q-Pharm Pty Ltd

IPD SHARING:
Plan to Share IPD: No